CLINICAL TRIAL: NCT07389655
Title: Mindful Awareness Practice (MAP) Pilot Randomized Controlled Trial for Older Adults With Mild Cognitive Impairment and Elevated Stress
Brief Title: (MAP) Pilot Randomized Controlled Trial for Older Adults With Mild Cognitive Impairment and Elevated Stress
Acronym: CohnMAP-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Ted K.S. Ng, Assistant Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 25093005
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment (MCI); Stress (Psychology)
Keywords: mindfulness; stress; MCI
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Awareness Practice (MAP) (Experimental): Mindful Awareness Practice (MAP)
  Interventions: Behavioral: Mindful Awareness Practice (MAP)
- Health Education Program (HEP) (Active Comparator): Health Education Program (HEP)
  Interventions: Behavioral: Mindful Awareness Practice (MAP)

INTERVENTIONS:
Behavioral: Mindful Awareness Practice (MAP) — Mindful Awareness Practice (MAP), a MBSR format-tailored to mild cognitive impairment (MCI)

SUMMARY:
The purpose of this study is to test whether a tailored mindfulness program, called the Mindful Awareness Practice (MAP) or a Health Education Program (HEP) can reduce stress and improve memory, mood, and well-being in older adults with Mild Cognitive Impairment (MCI) and elevated stress.

DETAILED DESCRIPTION:
The purpose of this study is to test whether a tailored mindfulness program, called the Mindful Awareness Practice (MAP) or a Health Education Program (HEP) can reduce stress and improve memory, mood, and well-being in older adults with Mild Cognitive Impairment (MCI) and elevated stress.

If you agree to participate in this study, your participation may last about 6 months, including 12 weeks of weekly sessions and 3 virtual/remotevisits (baseline, 3 months, 6 months).

You will be randomly assigned (like flipping a coin) to MAP mindfulness program or Health Education Program (HEP). Both programs involve 12 weeks of weekly 1-hour virtual sessions (recordings + some live Microsoft Teams). You will have 3 virtual/remote visits via phone or Microsoft Teams for cognitive testing, questionnaires, and to guide your self-collection of blood (finger-stick dried blood spot) and saliva samples. We will mail you the necessary collection kits in advance

There are risks to you for participating in this study. In this study, there is a very small risk that you may feel a little tired, frustrated or stressed especially during activities that involve thinking or answering questions; emotional discomfort during mindfulness activities; minor risks from finger stick dried blood spot collection, similar to checking blood sugar, which may include brief pain, mild bruising, or, very rarely, infection at the fingertip; and very small chance of loss of privacy of data despite strong safeguards. These risks are rare and we will do our best to prevent this from happening.

You may benefit from taking part in this study. Based on experience with mindful awareness program/health education program in patients with similar conditions, researchers believe it may be of benefit to people with your condition or it may be as good as standard therapy with fewer side effects. You may feel less stressed and have improved memory and mood. Even if you do not benefit directly, knowledge gained may help future programs to prevent Alzheimer's disease and related dementias. However, because individuals respond differently to interventions, no one can know in advance if it will be helpful for you.

ELIGIBILITY:
Inclusion Criteria:

* MCI participant: Community-dwelling, ≥65 years old, and diagnosed with MCI within the past 12 months, consented to participate in the trial, and have Wi-Fi access; Diagnosed with chronic stress-related conditions based on ICD-10 codes. No prior experience in mindfulness or other mind-body practices (e.g., yoga, Qi Gong, and Tai Chi) within the past year for >10 minutes per day28.

If taking medications with significant cholinergic, anticholinergic effects, anti-depressants, corticosteroid, or non-steroidal anti-inflammatory drug (NSAID), stabilized dose for ≥6 months.

* Ability to speak and read English
* Ability to provide informed consent

Exclusion Criteria:

* Diagnosed major psychiatric disorder, e.g., psychosis, bipolar disorder, and schizophrenia.Those with depression and anxiety will not be excluded, as they may be the prime targets for such an intervention and to avoid floor effects on measures that we suspected with our previous trial.

Diagnosed major neurological disorders, e.g., large vessel stroke, brain tumor, and severe brain injury.

Diagnosed terminal illness, including cancer, requiring palliative care, and organ failure, including hepatic or renal failure.

Sensory impairment, e.g., visual/hearing impairment impacting abilities to participate in the study.

Participating in other intervention(s) concurrently, either a research study or for self-interest (e.g., lifelong learning programs).which may improve memory for >2 days/week, 30 minutes a session in the past 3 months. After a wash-out period of ≥6 months, potential participants will be allowed to join this present study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Fidelity | From enrollment to the end of treatment at 12 weeks
  Rating of instructors will be done via 1) participant ratings using a softcopy delivery assessment form11 and 2) mindfulness-based interventions teaching assessment criteria scale13 to be filled up by the PI and co-I Krueger, viewing recordings of intervention sessions and comparing them against the a priori-designed intervention manuals.
Study Feasibility, including recruitment adherence and retention | From enrollment to the end of treatment at 12 weeks
  Recruitment = number of participants who consented to participate/number of potential participants who responded to recruitment/screened; Accrual & randomization = number of participants consented & passed eligibility criteria; goals: n=15 by recruitment month 3, n=25 by month 4.5, n=30 by month 5 or 6 (higher n at the beginning and tapering towards the end).
  Adherence = 1) the number of sessions attended at intervention 3-month & 6-month/total number of sessions offered (reasons for absence will also be noted for descriptive analyses and for informing future trial11), 2) the average number of minutes of: a. sessions attended and b. assigned homework completed by intervention 3-month & 6-month.
  Retention = 1) (of participants) the number of participants assessed at 3-month & 6-month /total number of participants randomized at baseline; 2) (of outcome measures) number of participants completed a specific outcome measure at 3-month & 6-month /total number of participants measured
Safety, indicated by number of adverse events | From enrollment to the end of treatment at 12 weeks
  The number of adverse events directly related to the delivery/receipt of the intervention10-12.
Acceptability (quantitative) | From enrollment to the end of treatment at12 weeks
  12-item adapted questionnaire used in a previous NIH-funded RCT14.The questions assess satisfaction with the intervention and perception of benefits conferred by the intervention11,15, such as: "Overall, how satisfied were participant with the MAP/HEP intervention?" "Did (& if so, how did) the intervention improve participant memory?" Similar to the original questionnaire11, each question has four options, i.e., "not at all", "a little", "some", and "a great deal". Acceptability will be based on the aggregate percentage of participants answering "some" and "a great deal", ranging from 0-100%.
Acceptability (qualitative) | From enrollment to the end of treatment at 12 weeks
  Measuring Acceptability (qualitative)

SECONDARY OUTCOMES:
Cognitive Outcomes | From enrollment to the end of treatment at12 weeks
  Boston story recall tests (attention, memory), Digit span forward & backward (memory, executive function), Category fluency (Fruits/Vegetables) (language), and 10-item MMSE (global cognition). Global Cognition Composite Score will be calculated based on the sum of z-scores of all tests. All tests are validated.
Depressive & anxiety symptoms | From enrollment to the end of treatment at12 weeks
  10-item CES-D and a 7-item Geriatric Anxiety Index (GAI).16 They are valid and have high reliability (α= 0.80 to 0.86 for CES-D and α= 0.85 to 0.92 for GAI).
Mindfulness | From enrollment to the end of treatment at12 weeks
  * Trait mindfulness: 15-item Five-facet Mindfulness Questionnaire (α=0.67 to 0.92)
  * State Mindfulness: 9-item Multidimensional State Mindfulness Questionnaire (MSMQ)(α=0.65-0.83)10617, (α=0.65-0.83 contingent on the facet/subscale).18
Perceived stress | From enrollment to the end of treatment at12 weeks
  10-item Perceived Stress Scale,19 an assessment of one's global appraisal of stress. The PSS has established validity and reliability (α=0.82).19
Social (dis) connections | From enrollment to the end of treatment at 12 weeks
  10-item UCLA Loneliness Scale; 7-item Positive Relations with Others sub-scale from the 42-item Ryff's Psychological Well-being Scale
Stress-related biomarker (Salivary cortisol) | From enrollment to the end of treatment at 12 weeks
  Measuring Stress-related biomarker (Salivary cortisol)
Dried blood spot (DBS) inflammatory and Alzheimer's disease (AD) biomarkers | From enrollment to the end of treatment at 12 weeks
  Stress-related biomarker (Salivary cortisol) Dried blood spot (DBS) inflammatory and Alzheimer's disease (AD) biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Ted Ng, PhD, Principal Investigator — Rush University Medical Center

IPD SHARING:
Plan to Share IPD: No